CLINICAL TRIAL: NCT04571736
Title: Interest of Improving Preoperative Medical Information by Video Support and Personalized and Secure Web Platform: Pilot Study in Thyroid Surgery (AMEDOP)
Brief Title: Pilot Study for Thyroid Surgery by Preoperative Video Support and Personalized and Secure Web Platform
Acronym: AMEDOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL19_0085 (7782); 2019-A02241-56 (Other: IDRCB)
Record Dates: First submitted 2020-07-27; First posted 2020-10-01 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Thyroid
Keywords: Preoperative Procedure; Instructional Films and Video
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- access to the internet information platform (Active Comparator): usual preoperative information and access to the internet information platform
  Interventions: Other: access to the internet information platform
- usual preoperative information (No Intervention): medical information delivered to the patient before any surgery

INTERVENTIONS:
Other: access to the internet information platform — This platform contains, among other things, an explanatory video of thyroid surgery and allows the patient to have access to information on surgical management at any time.
  Arms: access to the internet information platform

SUMMARY:
The medical information delivered to the patient before any surgery constitutes an essential and compulsory step during the initial management of the operated patient.

There are different reasons for the quantity and quality of medical information retained by the patient. An internet platform with personalized and secure access has been developed. This platform contains, among other things, an explanatory video of thyroid surgery and allows the patient to have access to information on surgical management at any time.

The investigators believe that unlimited access for the duration of the study to this platform could reduce the preoperative anxiety level of patients.

DETAILED DESCRIPTION:
The objective is to assess the impact of additional, personalized and accessible preoperative medical information via a secure internet platform on the anxiety level of patients before their surgery. For this, patients agreeing to participate in the study will be randomized (drawn at random) during the inclusion visit and divided into one of the following two groups:

* The control group: patients included in this group will receive the usual medical information as part of the surgery performed;
* The experimental group: the patients included in this group will have, in addition to the usual medical information, personalized and secure access to a platform so that they can have additional information on the surgery performed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75,
* Indication of lobo-isthmectomy or total thyroidectomy
* Compliance for the completion of self-questionnaires
* Person affiliated or beneficiary of a social security scheme.
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Difficulty understanding the French language
* Lack of internet access
* Persons placed under the protection of justice,
* Person under guardianship or curatorship
* Person participating in another research including an exclusion period still in progress,
* Subject with severely impaired physical and / or psychological health, which, according to the investigator, may affect the compliance of the study participant
* Pregnant / lactating woman

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2026-11-18 (Estimated); Study Completion 2027-03-18 (Estimated)

PRIMARY OUTCOMES:
Amsterdam Preoperative Anxiety and Information Scale (APAIS) SCORE | Baseline Day [-90 / -7] and Surgery Day [-1 / 0]
  rate of patients with perioperative anxiety symptoms refind by APAIS SCORE >= 11.
  Rate from 1 (absent) to 5 (extrem). Score 2 to 4 : rejection of information, 5 to 7 : medium desire for information, > 7 : hungry for information.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI-ETAT) SCORE | Baseline Day[ -90 / -7], Surgery Day [-1 / 0], discharge from the hospital Day [0 / 7] and postoperative visit Day [5-30]
  overall anxiety score. 20 items in the form of a 4-response Likert scale (from 1 : low anxiety to 4 : highest anxiety). The score goes from 20 to 80 depending of the degree of anxiety.
Internet use self-questionnaire | Baseline Day [-90 / -7]
  Description of internet use and median number of internet use during the preoperative period collected using the follow-up book given to the patient during the inclusion visit.
  4 items, if the answer for the 1st item is YES (Do you regulary consult the Internet for your health?) the subject must complete the item 2 and 4. If it's NO the subject must complete only the item 3.
  Item 2 is "why are you consulting internet" the subject had 3 possibility multiple choice questionnaire by answering with yes or no.
  Item 3 "Why the subject Don't use internet" 3 possibility multiple choice questionnaire by answering with yes or no.
  Item 4 "utility of the information found on internet" rate from 1 (none) to 5 (very important).
Internet use self-questionnaire | Surgery Day [ -1 / 0], Discharge from hospital Day [0-7] and postoperative visit Day [5-30]
  Description of internet use and median number of internet use during the preoperative period collected using the follow-up book given to the patient during post opérative visit.
  4 items, if the answer for the 1st item is YES (Do you regulary consult the Internet for your health?) the subject must complete the item 2 and 4. If it's NO the subject must complete only the item 3.
  Item 2 is "why are you consulting internet" the subject had 3 possibility multiple choice questionnaire by answering with yes or no.
  Item 3 "Why the subject Don't use internet" 3 possibility multiple choice questionnaire by answering with yes or no.
  Item 4 "utility of the information found on internet" rate from 1 (none) to 5 (very important).
specific questionnaire EDOP | post-operative visit Day [5-30] after viewing the screening video
  specific questionnaire in experimental group on the internet platform. 6 Items. Items 1, 2, 3, 6 in the form of a 5-response Likert scale (from 1: not satisfied at all, to 5 very satisfied).
  Item 4 number of times the platform is consulted. Item 5 is if the subject had consulted other website after consulting EDOP platform. If yes how many times, and the name(s) of the website, why did you consult website.
satisfaction assessment questionnaire and understanding of the preoperative medical information for control group | Baseline Day [-90 / -7], Surgery Day [-1/0], at discharge from hospital Day [0-7] and at the postoperative visit Day [5-30]
  Level of satisfaction and understanding obtained on the satisfaction assessment questionnaire and understanding of the preoperative medical information received for the control group.
  4 Items. Item 1 "quality of information" : 2 questions clear information and understanding in the form of a 5-response Likert scale (from 1: not at all, to 5 Totally).
  Item 2 necessity of complementary information, choice between no, a few, many information.
  Item 3 "comprehension on different topics explained by the physician conserning the surgery. This item is devided in 6 questions in the form of a 5-response Likert scale (from 1: not at all, to 5 Totally).
  Item 4 Visual analog scale rate from 0 not satisfied at all, to 100 totally satisfied.
satisfaction assessment questionnaire and understanding of the preoperative medical information for experimental groupe | 2 times at Baseline Day [-90 / -7] before and after the presentation of EDOP platform, Surgery Day [-1/0], at discharge from hospital Day [0-7] and at the postoperative visit Day [5-30]
  Level of satisfaction and understanding obtained on the satisfaction assessment questionnaire and understanding of the preoperative medical information received for experimental groupe before and after the presentation of the EDOP plateform.
  4 Items. Item 1 "quality of information" : 2 questions clear information and understanding in the form of a 5-response Likert scale (from 1: not at all, to 5 Totally).
  Item 2 necessity of complementary information, choice between no, a few, many information.
  Item 3 "comprehension on different topics explained by the physician conserning the surgery. This item is devided in 6 questions in the form of a 5-response Likert scale (from 1: not at all, to 5 Totally).
  Item 4 Visual analog scale rate from 0 not satisfied at all, to 100 totally satisfied.
State-Trait Anxiety Inventory (STAI-TRAIT) SCORE | Baseline Day[ -90 / -7]
  trait anxiety score. 20 items in the form of a 4-response Likert scale (from 1 : low anxiety to 4 : highest anxiety). The score goes from 20 to 80 depending of the degree of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Cartier, PI, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU Gui de Chauliac, Montpellier, Hérault, France